CLINICAL TRIAL: NCT02284100
Title: Animal-assisted Therapy in Pediatric Surgery: Cardiovascular, Neurological and Endocrinological Responses to Stress and Pain in the Immediate Post-operative Period
Brief Title: Animal-assisted Therapy in Pediatric Surgery: Post-operative Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Pelizzo Gloria, Professor, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20130005132
Record Dates: First submitted 2014-10-29; First posted 2014-11-05 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Surgery
MeSH Terms: interventions — Animal Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- animal assisted therapy group (Experimental): the dog was present during post-operative awakening (2 hours after surgery)
  Interventions: Behavioral: animal assisted therapy
- standard group (No Intervention): children had standard post-operative medical care

INTERVENTIONS:
Behavioral: animal assisted therapy — For the AAT session, a 7 year old Golden Retriever was employed as the therapy animal. Prior to the study, the dog underwent rigorous screening although she had previous experience in Animal Assisted Interventions and was already trained and prepared prior for this type of work. The dog was fully vaccinated, bathed regularly, screened for enteric pathogens, and treated for internal and external parasites on a monthly basis. The dog and handler met hospital policy for participating in animal-assisted therapy, including documentation of the dog's current vaccinations, controllability and temperament.
  The welfare of the dog was monitored and certificated by a dedicated veterinary during and at the end of the all sessions.
  Arms: animal assisted therapy group

SUMMARY:
The relationship between human beings and animals, especially dogs, has existed for thousands of years. Historically, animals have held an important role in this relationship as they provide company, stimulus and motivation. Animals are excellent company, since their visitation they do not discriminate or segregate any person, that is, they are free of prejudice.

In spite of the long-lasting presence of companion animals in human life, the idea that interaction with animals may exert a positive effect on human health is rather recent.

The American Veterinary Medical Association classifies therapeutic animal assisted interventions (AAI) into three categories: animal assisted activities (AAA) that utilize companion animals; animal assisted therapy (AAT) that utilizes therapy animals and service animal programs (SAP) that utilize service animals. AAT in particular, is a goal-directed intervention in which an animal that meets specific criteria is an integral part of the treatment process. AAT is technically defined as the use of trained animals by trained health professionals to facilitate specific, measurable goals for individual patients for whom there is documentation of progress .

Interest in AAT has been fueled by studies supporting the many health benefits. AAT has proven a useful adjunct in a variety of settings including mental health facilities, nursing homes and hospitals where most studies have been performed with adult patients with variable interventions, goals, patient characteristic and patient needs. In these studies, AAT resulted in significant reductions in anxiety, agitation and fear. In children, AAT dogs decreased distress during painful medical procedures, promoted calmness in children with post-traumatic stress disorders and increased attention and positive behaviors in children with pervasive developmental disorders.

Surgical procedures and hospitalization can be stressful for both children and their parents and they are associated with pain, helplessness, fear and boredom. AAT has been shown to facilitate a child's ability to cope with hospitalization, but to date, no studies on AAT benefits in pediatric surgery have been reported.

The purpose of this study was to better understand the effects of an AAT program on neurological, cardiovascular and endocrinological responses to stress and pain in the immediate post-operative period in children undergoing surgical procedures.

DETAILED DESCRIPTION:
Interest in animal-assisted therapy has been fueled by studies supporting the many health benefits in the adult and pediatric age. The purpose of this study was to study the impact of an AAT program on cardiovascular, neurological and endocrinological responses to stress and pain in the immediate post-operative period following pediatric surgery.

Forty immunocompetent children undergoing surgical procedures (including orchidopexy, inguinal or umbilical hernia repair, circumcision, varicocele treatment) were sequentially enrolled.

This was a randomised open-label, controlled, pilot study. The different arms consisted of an experimental group with a AAT session after a surgical procedure and a control group with standard care after surgery.

The study variables were determined in each patient independently of the assigned group, before and after the experimental intervention, by a researcher unblinded to the patient's group.

The outcomes of the study were to define the impact of AAT on neurological, cardiovascular and endocrinological signs, in response to stress and pain in children undergoing surgical procedures.

As outcome measures the investigators considered:

* for neurological impact, the difference in the prevalence of beta (>14 Hz) electroencephalogram (EEG) activity between intervention and control group (20-23);
* for autonomic impact, the difference in blood pressure (BP) between intervention and control group;
* for cardiac impact, the difference in heart rate (HR) between intervention and control group;
* for respiratory impact, the difference in oxygen saturation (SpO2) between intervention and control group;
* for cerebral oxygenation, the difference in prefrontal oxygenation (HbO2) with near-infrared spectroscopy (NIRS) between intervention and control group;
* for endocrinological impact, the difference in salivary cortisol levels, between intervention and control group. The Wong-Baker Faces pain scale (FPS) was used to measure the child's self-reported pain.

At admission, auxological examination of the children included measurement of height, weight and body mass index. Height measurement was performed with patients in an upright position, without shoes, with their heels together, arms extended down the sides of the body and head positioned parallel to the floor. Weight was measured with the children barefooted and wearing light clothes, standing upright in the centre of the scale platform with their arms extended down the sides of the body. BMI was calculated as body weight in kilograms divided by body height squared in meters.

EEG activity, cerebral prefrontal oxygenation, heart rate, blood pressure, oxygen saturation, salivary cortisol levels, faces pain scale were considered as indicators of neurological, cardiovascular and endocrinological response to stress and pain.

Data collection was performed in the following phases:

* for all parameters, post-operatively baseline (T1), two hours after surgery at re-admission to the Unit. Pre dog-intervention in the AAT-group;
* for all parameters, in the twenty minutes following T1 (T2). During the dog-intervention in the AAT-group. For the STAND-group, the child was asked to sit quietly;
* only for salivary cortisol levels, between 11 pm and midnight (T3, the time when cortisol is normally at its lowest)

Vitals signs

HR, BP, SpO2, HbO2 were monitored (Dräger Primus ®) and recorded as follows:

* T1 (every 5 minutes, for 10 minutes. Mean values were used for the statistical analysis);
* T2 (every 5 minutes, for 20 minutes. Mean values were used for the statistical analysis).

Endocrinological parameters Salivary cortisol levels were measured at T1, after T2 and T3. The saliva samples were collected using a standardized salivette and frozen at -20° until analysis in the laboratory. After thawing, salivary fluids were centrifugated to precipitate mucins and cortisol was assayed in the supernatant with a solid-phase radioimmunoassay, wherein 125-I labeled cortisol competes for a fixed time with cortisol in the biological sample (The Coat-A-Count Cortisol, Siemens, Los Angeles, CA).

Pain response The faces pain scale was used to measure the child's self-reported pain at T1 and at the end of T2. This scale consisted of 6 cartoon faces with varying expressions ranging from very happy to very sad. The child rated the pain intensity on a scale, with point 0 being no pain and point 10 being the worst pain.

Analgesic treatment in the first 12 hours post-intervention was recorded.

Electroencephalogram Regarding the AAT-group patients, an EEG recording was obtained when the child was awake, 2 hours after surgery and before and during AAT intervention. In the STAND-group patients, and EEG recording was made 2 hours after surgery.

Any change in the normal physiological structure of the EEG, correlating the effect of the anaesthesia, post-operative stress of AAT intervention was recorded and monitored.

In both cases, the protocol included an EEG recording tasting about 20 minutes, while awake, with open and closed eyes.

Parental permission was obtained through a written and oral informed consent. Written assent by the patient was also obtained in children eight years of age and older before enrolment.

Statistical analysis A desired sample size of 20 patients per group for a total of 40 subjects was determined based on 80% power alpha=0.10 (pilot study), using a 2-tailed test, to detect an effect size of 0.8 for the primary endpoint measured on a continuous scale, and an absolute difference in prevalence of the primary endpoint of 31 to 34% for the expected prevalence in the control group of 5 and 10% respectively.

Continuous variables were described as the mean and standard deviation (SD) or median and quartiles and categorical variables as counts and percentages. The prevalence of EEG beta activity was compared with the Fisher exact test. To test the effects of AAT on vital signs and on endocrinological parameters over time in the two groups, regression models for repeated measures were used, including a main effect for group and time, as well as their interaction. Distribution of pain scores at the end of the session in the two groups was compared with the Fisher exact test. A 2-sided p-value<0.05 was considered statistically significant. All statistical analyses were performed using Stata 13.1 (StataCorp, College Station, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* immunocompetent children (both genders)
* aged 3 to 17 years
* undergoing surgical procedures (including orchidopexy, inguinal or umbilical hernia repair, circumcision, varicocele treatment)

Exclusion Criteria:

* allergy or fear of dogs
* previous AAT experience
* immunodeficiency
* chronic illness
* obesity and use of any medications.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Neurological impact | Partecipants will be followed for the duration of immediate postoperative period, an expected average of 4 hours
  Neurological impact assessed by the difference in prevalence of beta (>14 Hz) electroencephalogram (EEG) activity between intervention and control group.

SECONDARY OUTCOMES:
Autonomic impact | Partecipants will be followed for the duration of immediate postoperative period, an expected average of 4 hours
  Autonomic impact assessed by the difference in blood pressure (BP) between intervention and control group
Cardiac impact | Partecipants will be followed for the duration of immediate postoperative period, an expected average of 4 hours
  Cardiac impact assessed by the difference in heart rate between intervention and control group
Respiratory impact | Partecipants will be followed for the duration of immediate postoperative period, an expected average of 4 hours
  Respiratory impact assessed by the difference in oxygen saturation (SpO2) between intervention and control group
Cerebral oxygenation | Partecipants will be followed for the duration of immediate postoperative period, an expected average of 4 hours
  Cerebral oxygenation assessed by the difference in prefrontal oxygenation (HbO2) between intervention and control group

OTHER OUTCOMES:
Endocrinological impact | Partecipants will be followed for the duration of immediate postoperative period, an expected average of 4 hours
  Endocrinological impact assessed by the difference in salivary cortisol levels between intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Pelizzo, Prof, Principal Investigator — Fondazione IRCCS Policlinico S. Matteo

REFERENCES:
- [Derived] Calcaterra V, Veggiotti P, Palestrini C, De Giorgis V, Raschetti R, Tumminelli M, Mencherini S, Papotti F, Klersy C, Albertini R, Ostuni S, Pelizzo G. Post-operative benefits of animal-assisted therapy in pediatric surgery: a randomised study. PLoS One. 2015 Jun 3;10(6):e0125813. doi: 10.1371/journal.pone.0125813. eCollection 2015. PMID 26039494